CLINICAL TRIAL: NCT00035503
Title: Multicenter Trial For Patients With Acute Crohn's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IXR-201-19-166
Record Dates: First submitted 2002-05-03; First posted 2002-05-06 (Estimated); Last update posted 2021-12-08 (Actual); Status verified 2021-12

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — etiprednol dicloacetate

INTERVENTIONS:
Drug: etiprednol dicloacetate

SUMMARY:
The purpose of this study is to see if etiprednol dicloacetate is safe and effective for the treatment of acute Crohn's disease.

ELIGIBILITY:
* Must have active confirmed Crohn's disease with CDAI > 220 and < 400.
* Otherwise healthy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-01-31 (Actual); Primary Completion 2004-01-31 (Actual); Study Completion 2004-01-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (9):
  - Stuart Weisman, Palo Alto, California
  - University of Colorado Medical Center, Denver, Colorado
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Mark Lamet, Hollywood, Florida
  - Wayne Schonfeld, Hollywood, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - University of Chicago Hospital Medical Center, Chicago, Illinois
  - Gerald Dryden, Louisville, Kentucky
  - Richard MacDermott, Albany, New York
- Canada (2):
  - Hillary Steinhart, Toronto, Ontario
  - Gary Wild, Montreal, Quebec